CLINICAL TRIAL: NCT07263555
Title: Clinical Performance of Alkasite-Based Resin Versus Nanohybrid Composite Resin Restorations for Occlusal Carious Lesions in Primary Molars: A Randomized Clinical Trial
Brief Title: Clinical Performance of Alkasite-based Restorations in Children
Acronym: Restorations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yusra hashim Mohamed kheir khogali, Master's degree student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Alkasite filling and caries
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Alkasite-based Restorations; Nano-hybrid Resin Composite
Keywords: Alkasite-based Restorations; Cention N; Nano-hybrid resin composite; clinical performance; secordary caries; Children; Class I

STUDY DESIGN:
Intervention Model Description: The included children with class I cavity carious lesions will be assigned to either alkasite-based restoration (Intervention group) or Nano-hybrid resin composite (Comparison group)
Who Masked: Participant, Outcomes Assessor
Masking Description: The children, outcome assessors, and the statistician will be blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alkasite-based Restorations (Cention N) (Experimental): The children assigned to this intervention group will have alkasite-based restorations for the treatment of Class I carious lesion in primary molars.
  Interventions: Other: Alkasite-based composite restorations
- Nano-hybrid composite resin restoration (TPH Spectra ST Universal Composite). (Active Comparator): The children assigned to the comparator group will undergo class I cavity restorations using nano-hybrid resin composite
  Interventions: Other: Nano-hybrid resin composite

INTERVENTIONS:
Other: Alkasite-based composite restorations — Alkasite-based restorations will be used in the treatment of class I carious lesion in primary molars.
  Other Names: Cention N
  Arms: Alkasite-based Restorations (Cention N)
Other: Nano-hybrid resin composite — Nanohybrid composite will be used in the restoration of Class I carious lesions in primary molars.
  Arms: Nano-hybrid composite resin restoration (TPH Spectra ST Universal Composite).

SUMMARY:
The aim of this study is to evaluate and compare the clinical performance of alkasite-based resin and nanohybrid composite resin materials in the restoration of occlusal carious lesions in primary molars of children.

DETAILED DESCRIPTION:
This randomized clinical trial aims to evaluate and compare the clinical performance of an alkasite-based resin restorative material (Cention N®) and a nanohybrid composite resin (TPH Spectra ST Universal Composite) in restoring occlusal carious lesions (Class I) in primary molars among children aged 4-6 years. Participants will be randomly allocated in a 1:1 ratio into two parallel groups and followed for a period of 12 months. The primary outcome will be the incidence of secondary caries assessed at 3, 6, and 12 months using the United States Public Health Service (USPHS) criteria, which grades restorations from Alpha (ideal/excellent) to Delta (failure). Secondary outcomes will include the evaluation of restoration fracture, marginal adaptation, marginal discoloration, surface roughness, and retention, all assessed at the same intervals using the same USPHS criteria.

ELIGIBILITY:
Inclusion Criteria:

* • Children aged 4-6 years of both sexes.

  * Cooperative children.
  * Apparently medically fit children according to parental history.
  * Children whose parents agree to sign the informed consent.
  * Children whose parents will be able to attend the follow-up.

Teeth:

* Primary molars with occlusal carious lesions (Class I), indicated for direct restorations.
* Teeth without signs of pulpal involvement, abscess, or fractures.

Exclusion Criteria:

Children:

* Children with systemic or mental disorders.
* Children whose parents refused to sign the informed consent.
* Noncompliant parent.
* Uncooperative children.

Teeth:

* Teeth with deep caries involving the pulp or clinical signs of pulpal infection (e.g., swelling, sinus, fistula, pathological mobility).
* Teeth with periapical pathology, internal or external root resorption, or mobility.
* Non-restorable teeth or lacking sufficient structure for restoration

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of secondary caries | 12 months
  The primary outcome of this study will be the evaluation of secondary caries incidence at 3, 6, and 12 months following restoration. Assessment will be carried out using the United States Public Health Service (USPHS) criteria, with restorations scored on a scale ranging from Alpha (clinically excellent) to Delta (clinically unacceptable.
  Each restoration will be scored as Alpha (A) if there is no evidence of secondary caries and the tooth-restoration interface remains intact. A score of Bravo (B) will indicate a questionable or suspicious area, such as slight marginal staining without definite cavitation. Charlie (C) will be assigned when definite secondary caries are observed, including softness or cavitation at the restoration margin, necessitating replacement of the restoration. Delta (D) will be used for severe carious lesions extending beneath the restoration, requiring immediate intervention.

SECONDARY OUTCOMES:
clinical evaluation of restoration fracture | 12 months
  The secondary outcomes will include the clinical evaluation of restoration fracture at 3, 6, and 12 months. The occurrence of restoration fracture will be evaluated using the United States Public Health Service (USPHS) criteria. Each restoration will be scored as Alpha (A) if no fracture is present and the restoration remains intact. A score of Bravo (B) will indicate minor chipping or superficial fracture that does not compromise function. Charlie (C) will be assigned when a fracture is evident that affects the integrity or function of the restoration, necessitating repair or replacement. Delta (D) will be used for severe fracture resulting in complete loss of the restoration, requiring immediate replacement.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Not determined yet.

REFERENCES:
- [Background] Attia, R., Sabry, R., Elafefy, A., & Essa, M. (2022). Clinical Performance of Alkasite Dental Material and High Viscosity Glass Ionomer Restorations in Class I Cavities. Comparative Study for One Year Follow Up. Egyptian Dental Journal, 68(4), 3881-3894.
- [Result] Arora D, Jain M, Suma Sogi HP, Shahi P, Gupta I, Sandhu M. In vivo evaluation of clinical performance of Cention N and glass ionomer cement in proximal restorations of primary molars. J Indian Soc Pedod Prev Dent. 2022 Jan-Mar;40(1):23-29. doi: 10.4103/jisppd.jisppd_108_21. PMID 35439879